CLINICAL TRIAL: NCT02093065
Title: Decreased Platelet Function as a Cause of Increased Bleeding in Patients With Hemophilia A
Brief Title: Platelet Function in Patients With Hemophilia A
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Alan D. Michelson, Professor of Pediatrics and Professor of Medicine, Harvard Medical School Director, Center for Platelet Research Studies Director, Thrombosis and Anticoagulation Program Boston Children's Hospital / Dana-Farber Cancer Institute, Boston Children's Hospital
Other Study IDs: BCH-CPRS-hemophilia A
Record Dates: First submitted 2014-03-19; First posted 2014-03-20 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Hemophilia A
Keywords: severe hemophilia A; coated platelets; bleeding
MeSH Terms: conditions — Hemophilia A; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Abnormalities in the gene encoding Factor VIII (FVIII) results in hemophilia A, an X-linked recessive bleeding disorder with a prevalence of 1 in 5000 males. Hemophilia A patients are classified into 3 different categories based on residual FVIII activity compared to normal: mild (6-40%), moderate (1-5%) and severe (<1%). This categorization correlates to some degree with bleeding phenotype, but does not completely define it. Some patients with hemophilia A bleed less often than others despite identical plasma FVIII levels. The cause(s) of this phenotype heterogeneity in hemophilia A remains largely unknown, despite a number of studies of possible factors.

Activated platelets, in addition to their role in primary hemostasis, play a major role in secondary hemostasis (coagulation) by providing a phospholipid surface to which coagulation factors bind. A role for platelets in the hemorrhagic propensity of hemophilia A has been suggested in the past, but only a small number of studies have been performed with limitations in assays performed and numbers of patients. The purpose of the present study is to determine whether platelet reactivity in severe hemophilia A patients is associated with past bleeding frequency and/or predicts future bleeding frequency.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe hemophilia A who are being prophylactically treated with FVIII.
* Age of at least 2 years.
* Bleeding history of at least 6 months.
* IRB-approved informed consent.

Exclusion Criteria:

* Presence of FVIII inhibitors.
* Greater than 7 days since active bleeding.

Ages: 2 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with severe hemophilia A who do not have inhibitors against FVIII and who have a bleeding history of at least 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2015-03; Primary Completion 2018-06 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
The percentage of coated platelets. | 2 years

SECONDARY OUTCOMES:
Platelet reactivity. | 2 years
The number of procoagulant platelet-derived microparticles. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alan D Michelson, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston Hemophilia Center, Boston, Massachusetts, United States